CLINICAL TRIAL: NCT04111575
Title: The Effect of Turkish Classical Music on Postpartum Pain and Anxiety in Women Who Delivered Via Cesarean Section
Brief Title: Music Therapy for Women, Delivered Via Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Eylem Toker, Assistant Professor Doctor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19.04.2017/No:7-35
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cesarean Section; Postpartum Period
Keywords: cesarean section; Music therapy; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Design, setting and subjects: The randomized controlled trial was conducted on 126 women who delivered via cesarean section in a tertiary hospital. The subjects were allocated to three groups (n=42 each) Interventions: In the experimental group 1 (once a day) and group 2 (twice a day) were made to listen to music for 30 minutes for two consecutive days. The control group routine care of 30 min a day in bed rest. The Personal Information Form, Visual Analog Scale, State-Trait Anxiety Inventory were administered to participants.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- music therapy group 1 (Experimental): The mothers in the experimental group 1 received music therapy for 30 minutes a day.They listened music for two consecutive days, considering the first day after the C-section as the beginning day.
  Interventions: Behavioral: Music Therapy
- music therapy group 2 (Experimental): The mothers in the experimental group 1 received music therapy for 30 minutes twice a day. They listened music for two consecutive days, considering the first day after the C-section as the beginning day.
  Interventions: Behavioral: Music Therapy
- control group (No Intervention): the control group were made to rest in bed for 30 minutes a day for two consecutive days, considering the first day after the C-section as the beginning day.

INTERVENTIONS:
Behavioral: Music Therapy — Music Therapy
  Other Names: musicotherapy
  Arms: music therapy group 1; music therapy group 2

SUMMARY:
Musical therapy is a type of therapy which is performed under a regular method by adjusting the physiological and psychological effects of musical tones and melodies in accordance with various situations. Therefore, the study was carried out as a randomized controlled trial in order to evaluate the effect of music therapy on the level of pain and anxiety in the postpartum period in women who delivered via cesarean section.

DETAILED DESCRIPTION:
Objectives: The study was carried out in order to determine the effect of music therapy on the level of postpartum pain and anxiety in women who delivered via cesarean section.

Design, setting and subjects: The randomized controlled trial was conducted on 126 women who delivered via cesarean section in a tertiary hospital. The subjects were allocated to three groups (n=42 each) Interventions: In the experimental group 1 (once a day) and group 2 (twice a day) were made to listen to music for 30 minutes for two consecutive days. The control group routine care of 30 min a day in bed rest. The Personal Information Form, Visual Analog Scale, State-Trait Anxiety Inventory were administered to participants. In the analysis of the data, one-way ANOVA, paired t-test, Kruskal Wallis-H and Wilcoxon tests were used.

Main outcome measures: State anxiety level and pain level.

ELIGIBILITY:
Inclusion Criteria:

* being at the age of 18 and above,
* being healthy,
* having given a live birth,
* having no hearing impairment,
* complication not having developed either in the mother or the baby

Exclusion Criteria:

* being at the age of 17 and below,
* being unhealthy,
* having given a stillbirth,
* having hearing impairment,
* complication having developed either in the mother or the baby

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | On the first and second days after C-section, change from first anxiety level at 30 minutes.The inventory has a Likert type scale of 20 items which aim to measure the state anxiety level.Higher scores indicate greater anxiety
  Anxiety level by State-Trait Anxiety Inventory
Visual Analog Scale (VAS) | On the first and second days after C-section, change from first pain level at 30 minute.The patient marks the pain he/she feels on a scale of 10 cm (100 mm), pain point 1 means "no pain", pain point 10 means "worst pain possible."
  Pain Level by Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Eylem TOKER, Kahramanmaraş, Dulkadiroglu, Turkey (Türkiye)

REFERENCES:
- [Background] Wu J, Chaplin W, Amico J, Butler M, Ojie MJ, Hennedy D, Clemow L. Music for surgical abortion care study: a randomized controlled pilot study. Contraception. 2012 May;85(5):496-502. doi: 10.1016/j.contraception.2011.09.018. Epub 2011 Nov 12. PMID 22079604
- [Background] Bally K, Campbell D, Chesnick K, Tranmer JE. Effects of patient-controlled music therapy during coronary angiography on procedural pain and anxiety distress syndrome. Crit Care Nurse. 2003 Apr;23(2):50-8. No abstract available. PMID 12725195
- [Background] Ebneshahidi A, Mohseni M. The effect of patient-selected music on early postoperative pain, anxiety, and hemodynamic profile in cesarean section surgery. J Altern Complement Med. 2008 Sep;14(7):827-31. doi: 10.1089/acm.2007.0752. PMID 18803492
- [Background] Tournaire M, Theau-Yonneau A. Complementary and alternative approaches to pain relief during labor. Evid Based Complement Alternat Med. 2007 Dec;4(4):409-17. doi: 10.1093/ecam/nem012. PMID 18227907
- [Background] Toker E, Komurcu N. Effect of Turkish classical music on prenatal anxiety and satisfaction: A randomized controlled trial in pregnant women with pre-eclampsia. Complement Ther Med. 2017 Feb;30:1-9. doi: 10.1016/j.ctim.2016.11.005. Epub 2016 Nov 18. PMID 28137517
- [Background] Bekiroglu T, Ovayolu N, Ergun Y, Ekerbicer HC. Effect of Turkish classical music on blood pressure: a randomized controlled trial in hypertensive elderly patients. Complement Ther Med. 2013 Jun;21(3):147-54. doi: 10.1016/j.ctim.2013.03.005. Epub 2013 Apr 2. PMID 23642944
- [Background] Shin HS, Kim JH. Music Therapy on Anxiety, Stress and Maternal-fetal Attachment in Pregnant Women During Transvaginal Ultrasound. Asian Nurs Res (Korean Soc Nurs Sci). 2011 Mar;5(1):19-27. doi: 10.1016/S1976-1317(11)60010-8. Epub 2011 Apr 5. PMID 25029946
- [Background] Laopaiboon M, Lumbiganon P, Martis R, Vatanasapt P, Somjaivong B. Music during caesarean section under regional anaesthesia for improving maternal and infant outcomes. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD006914. doi: 10.1002/14651858.CD006914.pub2. PMID 19370660
- [Background] Handan E, Sahiner NC, Bal MD, Dissiz M. Effects of Music during Multiple Cesarean Section Delivery. J Coll Physicians Surg Pak. 2018 Mar;28(3):247-249. doi: 10.29271/jcpsp.2018.03.247. PMID 29544589
- [Background] Hepp P, Hagenbeck C, Gilles J, Wolf OT, Goertz W, Janni W, Balan P, Fleisch M, Fehm T, Schaal NK. Effects of music intervention during caesarean delivery on anxiety and stress of the mother a controlled, randomised study. BMC Pregnancy Childbirth. 2018 Nov 3;18(1):435. doi: 10.1186/s12884-018-2069-6. PMID 30390639
- [Background] Moradipanah F, Mohammadi E, Mohammadil AZ. Effect of music on anxiety, stress, and depression levels in patients undergoing coronary angiography. East Mediterr Health J. 2009 May-Jun;15(3):639-47. PMID 19731780
- [Background] Ferrer AJ. The effect of live music on decreasing anxiety in patients undergoing chemotherapy treatment. J Music Ther. 2007 Fall;44(3):242-55. doi: 10.1093/jmt/44.3.242. PMID 17645387
- [Background] Tseng YF, Chen CH, Lee CS. Effects of listening to music on postpartum stress and anxiety levels. J Clin Nurs. 2010 Apr;19(7-8):1049-55. doi: 10.1111/j.1365-2702.2009.02998.x. PMID 20492049
- [Background] Kafali H, Derbent A, Keskin E, Simavli S, Gozdemir E. Effect of maternal anxiety and music on fetal movements and fetal heart rate patterns. J Matern Fetal Neonatal Med. 2011 Mar;24(3):461-4. doi: 10.3109/14767058.2010.501122. Epub 2010 Jul 7. PMID 20608798
- [Background] Yang M, Li L, Zhu H, Alexander IM, Liu S, Zhou W, Ren X. Music therapy to relieve anxiety in pregnant women on bedrest: a randomized, controlled trial. MCN Am J Matern Child Nurs. 2009 Sep-Oct;34(5):316-23. doi: 10.1097/01.NMC.0000360425.52228.95. PMID 19713801
- [Background] Vianna MN, Barbosa AP, Carvalhaes AS, Cunha AJ. Music therapy may increase breastfeeding rates among mothers of premature newborns: a randomized controlled trial. J Pediatr (Rio J). 2011 May-Jun 8;87(3):206-12. doi: 10.2223/JPED.2086. Epub 2011 Apr 1. English, Portuguese. PMID 21461451
- [Background] Lai HL, Chen CJ, Peng TC, Chang FM, Hsieh ML, Huang HY, Chang SC. Randomized controlled trial of music during kangaroo care on maternal state anxiety and preterm infants' responses. Int J Nurs Stud. 2006 Feb;43(2):139-46. doi: 10.1016/j.ijnurstu.2005.04.008. Epub 2005 Jul 5. PMID 15996669
- [Background] Whipple J. The effect of parent training in music and multimodal stimulation on parent-neonate interactions in the neonatal intensive care unit. J Music Ther. 2000 Winter;37(4):250-68. doi: 10.1093/jmt/37.4.250. PMID 11281808
- [Background] Kimber L, McNabb M, Mc Court C, Haines A, Brocklehurst P. Massage or music for pain relief in labour: a pilot randomised placebo controlled trial. Eur J Pain. 2008 Nov;12(8):961-9. doi: 10.1016/j.ejpain.2008.01.004. Epub 2008 Mar 4. PMID 18304848
- [Background] Bulfone T, Quattrin R, Zanotti R, Regattin L, Brusaferro S. Effectiveness of music therapy for anxiety reduction in women with breast cancer in chemotherapy treatment. Holist Nurs Pract. 2009 Jul-Aug;23(4):238-42. doi: 10.1097/HNP.0b013e3181aeceee. PMID 19574761
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Chang SC, Chen CH. Effects of music therapy on women's physiologic measures, anxiety, and satisfaction during cesarean delivery. Res Nurs Health. 2005 Dec;28(6):453-61. doi: 10.1002/nur.20102. PMID 16287051
- [Background] Lin HH, Chang YC, Chou HH, Chang CP, Huang MY, Liu SJ, Tsai CH, Lei WT, Yeh TL. Effect of music interventions on anxiety during labor: a systematic review and meta-analysis of randomized controlled trials. PeerJ. 2019 May 15;7:e6945. doi: 10.7717/peerj.6945. eCollection 2019. PMID 31143552
- [Background] Reza N, Ali SM, Saeed K, Abul-Qasim A, Reza TH. The impact of music on postoperative pain and anxiety following cesarean section. Middle East J Anaesthesiol. 2007 Oct;19(3):573-86. PMID 18044285
- [Background] Şahin, NH. Cesarean Section: Prevalence and Consequences. Journal of Maltepe University Nursing Science and Art 2009;2:93-98.
- [Background] Altuntaş H., Dansuk R., Köse O. Evaluation of Cesarean Ratios in Terms of Several Variables. KÜ Tıp Fak Derg 2013;15: 1-7.
- [Background] Yüksel N. Anxiety disorders. In: Yüksel N, ed. Mental Disorders. 3rd ed. Ankara:MN Medikal & Nobel; 2006:143-182.
- [Background] Gürkan A, Bilge A. Alternative therapies and psychiatric nursing. Ege Univ JNurs High School. 2006;22:225-232.
- [Background] Schmidt LA, Trainor LJ. Frontal brain electrical activity (EEG) distinguishes valence and intensity of musical emotions. Cogn Emot. 2001;15:487-500.
- [Background] Chlan L. A review of the evidence for music intervention to manage anxiety in critically ill patients receiving mechanical ventilatory support. Arch Psychiatr Nurs. 2009 Apr;23(2):177-9. doi: 10.1016/j.apnu.2008.12.005. PMID 19327560
- [Background] Wakim JH, Smith S, Guinn C. The efficacy of music therapy. J Perianesth Nurs. 2010 Aug;25(4):226-32. doi: 10.1016/j.jopan.2010.05.009. PMID 20656259
- [Background] Procelli DE. The effects of music therapy and relaxation prior to breastfeeding on the anxiety of new mothers and the behavior state of their ınfants during feeding. F.S.U. College of Music, MA Thesis, Florida, United States; 2005.
- [Background] Mamuk R, Davas Nİ. Non-pharmacological relaxation and sensual stimulation methods used in the control of delivery pain. Med Bull Sisli Etfal Hosp. 2010;44:137-144.
- [Background] Ersanlı C. The effect of music listened by primigravidae treated with induction of labor through training during labor on delivery process. M.U. Health Sciences Institute, MA Thesis, Istanbul, Turkey; 2007.
- [Background] Çatalgöl Ş. The effect of ney sound listened by primigravidae treated with induction of labor through training during labor on delivery process. E U. Health Sciences Institute, MA Thesis, İzmir; 2013
- [Result] Simavli S, Gumus I, Kaygusuz I, Yildirim M, Usluogullari B, Kafali H. Effect of music on labor pain relief, anxiety level and postpartum analgesic requirement: a randomized controlled clinical trial. Gynecol Obstet Invest. 2014;78(4):244-50. doi: 10.1159/000365085. Epub 2014 Sep 16. PMID 25227477
- See also: The World Health Statistics 2014. Accessed from: 2018 — http://apps.who.int/iris/bitstream/10665/112738/1/9789240692671_eng.pdf?ua=1.